CLINICAL TRIAL: NCT03719677
Title: Reducing Metabolic Syndrome and Unmet Needs Among Rural Breast Cancer Survivors During the Survivorship Transition
Brief Title: Reducing Metabolic Syndrome Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Heather Fritz, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-062
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habit development intervention (Experimental): Treatment includes occupational therapy evaluation and consultation to address any deficits in physical function, safety, social participation and/or life roles. After the occupational therapy evaluation, the therapist delivers education on physical activity and dietary recommendations and habit development techniques, and uses behavioral skills training to develop habit plans, as well as prompts/cues, environmental modifications, and reminder text messages to reinforce engagement in the plan. The intervention is delivered through 3 face to face sessions, 9 tele coaching calls, and text messages.
  Interventions: Behavioral: Habit development intervention

INTERVENTIONS:
Behavioral: Habit development intervention — Lifestyle behavior change intervention targeting physical activity and dietary habit development as well as improving physical and social functioning

SUMMARY:
Using a pilot 1-arm pre-post design, investigators will implement an intervention that is personalized, low burden (the majority of interactions are telephone coaching sessions), and delivered during the initial survivorship transition.

To determine the feasibility of the intervention 48 community-dwelling rural breast cancer survivors (BCS) (ages 40 and older) will receive the intervention. The 12-week intervention consists of three home-based face-to-face consultations with the therapist, 9 weekly habit tele phone coaching sessions, and the use of implementation intentions, environmental modifications, and tailored text messages to support physical activity and dietary habit formation and address unmet needs.

DETAILED DESCRIPTION:
The objective of the present study is to determine the feasibility of a manual, theory based, occupational therapist delivered, preventative intervention to increase habit development (HD) of healthy dietary and physical activity behaviors, and reduce metabolic syndrome (MetS) among high-risk, rural breast cancer survivors (BCS). Using a pilot 1-arm pre-post design, investigators will implement an intervention that is personalized, low burden (the majority of interactions are telephone coaching sessions), and delivered during the initial survivorship transition. To determine the feasibility of the intervention 48 community-dwelling rural BCS (ages 40 and older) will receive the intervention. The 12-week intervention consists of three home-based face-to-face consultations with the therapist, 9 weekly habit telephone coaching sessions, and the use of implementation intentions, environmental modifications, and tailored text messages to support physical activity and dietary habit formation and address unmet needs. Feasibility metrics will be collected throughout the intervention. The one specific aim is:

Aim 1. To determine the feasibility and acceptability of the intervention for rural BCS. Investigators will evaluate recruitment, trial engagement and retention rates, treatment satisfaction, and the feasibility of the data collection processes for the primary behavioral measures of HD.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Diagnosis of stage 1-3 histologically confirmed first cancer of the breast
* Reside in a zip code designated as rural by the United States Department of Agriculture Economic Research Service
* Be within the initial 12 months following the end of primary treatment and meet 3 of the following 5 criteria for MetS confirmed via point-of-care testing or documentation in their medical record:

A large waistline > 35 inches Blood pressure > 130/85; HbA1c of 5.7%-6.4%; Triglyceride levels > 150 mg/dL; HDL cholesterol levels < 50 mg/dL

Exclusion Criteria:

* Will not exclude participants based on hormone receptivity, one exception is that we will exclude HER2 positive BCS
* Pregnant patients
* Resistant Hypertension
* Steroid-dependent asthma or Chronic obstructive pulmonary disease
* Cirrhosis or hepatic failure
* A major cardiovascular event (e.g., stroke, myocardial infarction) within the previous 90 days
* Chronic kidney disease on renal replacement therapy
* Type one or two diabetes
* Stage 4 cancer; those with a secondary cancer (except for nonmelanomatous skin cancers and carcinoma of the cervix in situ)
* Taking weight loss medications
* Current involvement in a behavioral program
* Neuropsychiatric disorder or dementia

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Fritz, PhD, Principal Investigator — Wayne State University
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Habit Development Intervention
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Habit Development Intervention
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Behavioral Automaticity Index
Description: Measures changes in habit strength, scores range from 1-7 with higher scores indicating a stronger habit
Time Frame: From week 0-2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Habit Development Intervention
Number analyzed (Participants) | 7
score on a scale
  Baseline | 1.6 (1.3)
  Post test | 4.8 (2.1)

ADVERSE EVENTS:
Time Frame: 3 months
Description: The treatment involved providing education and counseling about how to develop healthy dietary and physical activity habits. No invasive procedures or hands on treatments or pharmacological agents were included in the study. There are no known risks for serious adverse events, or all cause mortality from health coaching interventions limited to diet and physical activity. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were monitored/assessed at each study visit.
Arm/Group | Habit Development Intervention
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03719677/Prot_SAP_000.pdf